CLINICAL TRIAL: NCT02593370
Title: Suprasacral Parallel Shift - Ultrasound/MR Image Fusion Guided Lumbosacral Plexus Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas F. Bendtsen (Other)
Collaborators: AP Moeller Foundation (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Thomas F. Bendtsen, Research anesthetist, ass. professor, PhD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AUH-TFB-SSPS
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Hip Fractures; Anesthesia Local; Pain, Perioperative
Keywords: Hip surgery anesthesia; Perioperative analgesia
MeSH Terms: conditions — Hip Fractures; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suprasacral Parallel Shift guided by US/MR image fusion (Experimental): Use of ultrasound/MR image fusion guided Suprasacral Parallel Shift technique to place a lumbar plexus block (20 mL 2% lidocaine with epinephrine added gadoterate meglumine).
  Interventions: Drug: Lidocaine-epinephrine added gadoterate meglumine
- Suprasacral Parallel Shift guided by US (Active Comparator): Use of ultrasound guided Suprasacral Parallel Shift technique to place a lumbar plexus block (20 mL 2% lidocaine with epinephrine added gadoterate meglumine).
  Interventions: Drug: Lidocaine-epinephrine added gadoterate meglumine

INTERVENTIONS:
Drug: Lidocaine-epinephrine added gadoterate meglumine

SUMMARY:
The main objective of the trial is to complete a double-blinded randomized controlled trial with crossover design of a lumbosacral plexus block with the Suprasacral Parallel Shift technique guided by ultrasound/magnetic resonance (MR) image fusion vs. Suprasacral Parallel Shift guided by ultrasound by estimating sensory block of the femoral nerve, the obturator nerve, the lumbosacral trunk, and spinal nerve L1 in healthy volunteers.

DETAILED DESCRIPTION:
The main objective of the trial is to complete a double-blinded randomized controlled trial with crossover design of a one-injection nerve block of the lower part of the lumbar plexus and the upper part of the sacral plexus (Suprasacral Parallel Shift, SSPS) to achieve analgesia of the femoral nerve, the obturator nerve, the lumbosacral trunk, and spinal nerve L1 with SSPS guided by ultrasound/MR image fusion vs. SSPS guided by ultrasound by estimating sensory block of in healthy volunteers by estimating the sensory block of dermatomes of the terminal nerves in healthy volunteers.

The secondary objective is to estimate a) preparation and b) procedure time, c) injection site and d) depth, e) discomfort, f) change in MAP, g) plasma lidocaine pharmacokinetics, h) motor and i) sensory block, j) perineural and k) epidural spread of lidocaine-epinephrine added gadotorate meglumine on MRI, and l) cost-effectiveness of SSPS guided by ultrasound/MR image fusion vs. SSPS guided by ultrasound.

The investigators hypothesize that block success is higher for SSPS guided by ultrasound/MR image fusion than for SSPS guided by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Volunteers who has given their written and oral informed consent to participate in the study after having fully understood the content and the limitations of the protocol.
* Normal healthy person (American Society of Anesthesiology [ASA] Classification I)

Exclusion Criteria:

* Volunteers not able to cooperate in the study
* Volunteers not able to understand or speak Danish
* Daily use of analgesics
* Allergy against the medicines used in the study
* Drug abuse (according to the investigator's judgement)
* Alcohol consumption greater than the recommendations of the Danish National Board of Health
* Contraindication for MRI including pregnancy
* Volunteer in whom nerve blocks are not possible due to technical reasons
* Volunteer who are incompetent (ie. surrogate consent is not accepted)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Block success | Estimated 40 min after completed intervention. Presented 10 months after last patient last visit (LVLP).
  Block success of the clinical relevant lumbosacral nerves that innervate the hip joint capsule estimated as significant motor block of the obturator nerve, the femoral nerve, and the lumbosacral trunk. Motor block is a significant proxy marker of sensory block. Motor block (muscle strength, mmHg) is assessed with a handheld dynamometer.

SECONDARY OUTCOMES:
Plasma lidocaine | Blood samples are withdrawn 0, 5, 10, 20, 40, 60, and 90 minutes after intervention. Presented 10 months after LVLP
Time for preparation | Estimated prior to intervention. Presented 10 months after LVLP
  Time for preparation in seconds is defined as the time of placement of the volunteer on the bed until the end of pre-ultrasound scanning
Block procedure time | Estimated during intervention. Presented 10 months after LVLP
  Block procedure time in seconds is defined as the time of the placement of the ultrasound probe on the skin to until the block needle is pulled out after injection of local anesthetics
Injection site | Estimated at the end of the intervention. Presented 10 months after LVLP
Block needle depth | Estimated at the end of the intervention. Presented 10 months after LVLP
Discomfort | Estimated immediately after the intervention. Presented 10 months after LVLP
  Estimated on numeric rating scale 0-10
Mean arterial pressure change | Mean arterial pressure is measured prior intervention and 5 min after intervention. Presented 10 months after LVLP
Sensory (cold, warm, touch, pain) block of the dermatomes T12-S3 and the lateral femoral cutaneous nerve | Estimated 50 min after intervention. Presented 10 months after LVLP
Perineural spread of local anesthetics added gadoterate meglumine | Estimated on MRI sampled 10-30 minutes after intervention. Presented 10 months after LVLP
Epidural spread of local anesthetics added gadoterate meglumine | Estimated on MRI sampled 10-30 minutes after intervention. Presented 10 months after LVLP
Cost-effectiveness (ICER) | Calculated after LVLP. Presented 10 months after the last visit of the last volunteer
  ICER is estimated as the difference in mean marginal cost of the blocks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Strid JM, Pedersen EM, Al-Karradi SN, Bendtsen MA, Bjorn S, Dam M, Daugaard M, Hansen MS, Linnet KD, Borglum J, Soballe K, Bendtsen TF. Real-Time Ultrasound/MRI Fusion for Suprasacral Parallel Shift Approach to Lumbosacral Plexus Blockade and Analysis of Injectate Spread: An Exploratory Randomized Controlled Trial. Biomed Res Int. 2017;2017:1873209. doi: 10.1155/2017/1873209. Epub 2017 Mar 15. PMID 28396863